CLINICAL TRIAL: NCT03373773
Title: Home vs. Office Foley Catheter Removal in Women With Voiding Difficulty Following Pelvic Reconstructive Surgery: A Randomized Controlled Trial
Brief Title: Home vs. Office Foley Catheter Removal in Women With Voiding Difficulty Following Pelvic Reconstructive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000030019; 2000022371 (Other: Old Yale HIC IRB #)
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Voiding Disorders
Keywords: pelvic reconstructive surgery; foley catheter; Foley removal; Urogynecology; Urinary Retention; Gynecologic surgery
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Home Removal (Active Comparator): Patients will be randomly allocated to two groups: subjects in one group will remove their indwelling Foley catheter at home and will have voiding assessment remotely based on their voiding characteristics (a Force of Stream of >5/10 indicates that the patient has adequate bladder function), and the other group will follow up in the office for Foley catheter removal and voiding trial.
  Subjects in this arm will remove the Foley catheter at home.
  Interventions: Procedure: Foley catheter removal
- Office Removal (Active Comparator): Patients will be randomly allocated to two groups: subjects in one group will remove their indwelling Foley catheter at home and will have voiding assessment remotely based on their voiding characteristics (a Force of Stream of >5/10 indicates that the patient has adequate bladder function), and the other group will follow up in the office for Foley catheter removal and voiding trial.
  Subjects in this arm will remove the Foley catheter in a medical office.
  Interventions: Procedure: Foley catheter removal

INTERVENTIONS:
Procedure: Foley catheter removal — After reinsertion of the Foley catheter, both groups of women will be given instructions on urinary catheter and bag management, this will be done by an RN as per standard protocol. Prior to discharge, every subject from the home removal group as well as their significant other/caregiver/family member will receive a standardized education session and written and illustrated instructions on Foley catheter removal from RN, per standard protocol. They will be provided with the syringe for catheter removal, urine collection pan, and a diary to record their voiding quality and quantity. Both groups of women will have the catheter removal in 2 days.

SUMMARY:
The purpose of this study is to evaluate the patient satisfaction with voiding assessment remotely after removal of Foley catheter at home by the patient or her caregiver compared to removal at the office by a healthcare provider in patients who have been diagnosed to have voiding difficulty after pelvic reconstructive surgery.

DETAILED DESCRIPTION:
While in the hospital, all women who undergo surgery for pelvic organ prolapse and/or urinary incontinence will have a voiding trial to evaluate whether their bladder is working as it should. A voiding trial is when you are asked to urinate when you feel the desire to do so, sometimes, a physician may fill your bladder with water prior to removing the Foley catheter. This allows the physician to know exactly how much is left in your bladder. This evaluation will occur in the recovery room for subjects who have a same-day procedure. Those who are admitted to the hospital will have the voiding trial before their discharge typically on postoperative day 1. Those who fail the voiding trial will be diagnosed with urinary retention (bladder not working as well as we expect) and will be discharged home with a Foley catheter. If you agree to participate you will be randomly assigned to one of two groups: Subjects in the one group will remove their indwelling Foley catheter at home and will have a voiding assessment done over the telephone based on their self-reported force of urinary stream. The other group will follow up in the Uro/Gynecology office for Foley catheter removal and voiding trial. Which group you are assigned to will be random. You have an equal chance to be assigned to either group. It is important to note that outside of the study, physicians choose to manage patients one of these two ways. Removal of the Foley catheter at home is not experimental, and often done in these situations.

Both groups of women will be given instructions on urinary catheter and bag (where the urine drains into) management. Prior to discharge, every subject from the home removal group as well as their significant other/caregiver/family member if applicable will receive a standardized education session and written and illustrated instructions on Foley catheter removal. This teaching will be done by an experienced and qualified nurse. You will be provided with the syringe for catheter removal, urine collection pan, and a diary to record their voiding quality and quantity. Both groups of women will have the catheter removal in 2 days. This will have to be delayed up to 4 days due to weekends if the procedure is performed on a Thursday or Friday.

In the home removal group, you and your significant other/caregiver/family member will be instructed to remove the Foley catheter at the pre-set date prior to 8 am. The research nurse or Uro/Gynecology (uro/Gyn) office nurse will contact contact 4 hours after removal. Voiding function will be evaluated by your self reported Force of Stream (FOS). This means the force that urine is expelled from your body compared to normal. A report of FOS of at least 5 on a 0-10 has been shown to be a safe and effective method of assessing voiding function. Additionally, volume of each void will be measured by you and reported to the research nurse and/or the UroGyn office nurse. If there is evidence of voiding difficulty as indicated by a FOS below 5/10, the research and/or UroGyn nurse will instruct you to follow up in the office immediately for clean intermittent self-catheterization (CISC) teaching. This means inserting a small, thin plastic tube in your urethra (opening of the body where urine is expelled). If your voiding pattern qualifies as adequate, you will not require an office visit for voiding assessment. However, you will be instructed to contact the office if you feel full after voiding, are voiding less than 2 ounces or 50 mL each time and more often than every 30 minutes, or feel pressure and discomfort in their lower abdomen.

Women in the other group will return to the office in 2-4 days and will undergo a voiding trial via retrograde fill with 10 ounces (300 mL) of normal saline or until your bladder capacity is reached. This means that a catheter will be inserted in your urethra and normal saline will be put in your bladder via a large syringe that acts as a funnel. You would be considered to have failed the voiding trial and be taught clean intermittent self-catheterization if you do not void 5 ounces (150 mL) within an hour or you become too uncomfortable with the bladder fullness, and your postvoid residual volume is greater than 150 mL. The residual volume is determined by a portable ultrasound like machine via an external probe which is scanned over your lower pelvic area.

At the routine 2 - 4 week post-operative visit, both groups will receive a 5 question survey asking about your experience with removal of the Foley catheter.

ELIGIBILITY:
Inclusion Criteria:

* Women with post-operative voiding difficulty requiring catheterization after pelvic reconstructive surgery or surgery for urinary incontinency.

Exclusion Criteria:

* A Pelvic Reconstructive Surgery/Urogynecology fellow or attending physician may deem patients ineligible based on patients post-operative voiding trial.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Up to 4 weeks
  At the routine 2-4 week post-operative visit, patients will be given an internally developed 5 item visual analogue scale regarding their experience with the Foley-catheter removal. The item used as the primary outcome measure will ask "How satisfied were you with the overall removal process of the Foley catheter?"
  Lower scores indicate less satisfaction, higher scores higher satisfaction.

SECONDARY OUTCOMES:
Removal Method Negative Emotions | Up to 4 weeks
  At the routine 2-4 week post-operative visit, patients will be given an internally developed 5 item visual analogue scale regarding their experience with the Foley-catheter removal. This item used asks "Did you experience any negative emotions during the removal process (e.g. fear, anxiety ect.)?"
  Lower scores indicate greater negative emotions, higher scores indicate fewer negative emotions.
Removal Method Recommendation | Up to 4 weeks
  At the routine 2-4 week post-operative visit, patients will be given an internally developed 5 item visual analogue scale regarding their experience with the Foley-catheter removal. This item used asks "How likely would you be to recommend your method of Foley catheter removal to a friend/family member, if they were in the same situation?"
  Lower scores indicate less likely to recommend, higher scores indicate more likely to recommend.
Removal Method Convenience | Up to 4 weeks
  At the routine 2-4 week post-operative visit, patients will be given an internally developed 5 item visual analogue scale regarding their experience with the Foley-catheter removal. This item used asks "How convenient was the process of Foley catheter removal (e.g. time, ease ect.)?"
  Lower scores indicate less convenient, higher scores indicate more convenient.
Removal Method Preference | Up to 4 weeks
  At the routine 2-4 week post-operative visit, patients will be given an internally developed 5 item visual analogue scale regarding their experience with the Foley-catheter removal. This item used asks "Where would you prefer your Foley catheter removed?"
  Lower scores indicate preference for office removal, higher scores indicate preference for home removal.

CONTACTS AND LOCATIONS:
Overall Officials: Oz Harmanli, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Popiel P, Getaneh F, Yeh J, Rickey L, Bercik R, Harmanli O. Voided Volume for Assessment of Bladder Emptying After Female Pelvic Floor Surgery: A Randomized Controlled Trial. Urogynecology (Phila). 2022 Dec 1;28(12):811-818. doi: 10.1097/SPV.0000000000001230. Epub 2022 Jun 22. PMID 36409638